CLINICAL TRIAL: NCT01203618
Title: Exploratory Phase 2 Study of Farletuzumab in Resectable Non-functioning Pituitary Adenoma
Brief Title: Exploratory Study of Farletuzumab to Treat Resectable, Non-functioning Pituitary Adenomas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated due to focus of primary therapeutic areas.
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAb-003-007
Record Dates: First submitted 2010-07-28; First posted 2010-09-16 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Resectable, Non-functioning Pituitary Adenoma
Keywords: Resectable, non-functioning pituitary adenoma; Pituitary tumor; Pituitary adenoma; Pituitary macroadenoma
MeSH Terms: conditions — Pituitary Neoplasms | interventions — farletuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Farletuzumab — Farletuzumab initial loading dose 5.0 mg/kg intravenous followed by 2.5 mg/kg intravenous for all subsequent doses every 2 weeks for up to 12 months.
  Other Names: MORAb-003

SUMMARY:
The purpose of this study is to evaluate whether therapy with farletuzumab is effective and safe in the treatment of resectable, non-functioning pituitary adenomas.

DETAILED DESCRIPTION:
Non-functioning pituitary adenomas are the most frequent type of pituitary tumors, defined by the lack of hormonal overproduction from the tumor. Non-functioning macroadenomas are > 1 cm in size that can cause progressive visual loss, headaches, and symptoms of pituitary dysfunction (hypopituitarism and/or hyperprolactinemia). Initial treatment for these type of tumors is trans sphenoidal surgical resection. In cases where the outcome is incomplete surgical resection of the tumor, repeat surgery and external beam radiation therapy may be performed. Previous clinical work suggests there may be a role for a folate receptor in the treatment of non-secretory, pituitary adenomas. MORAb-003 is a monoclonal antibody that has the potential to be an effective agent against resectable, non-functioning pituitary adenomas. MORAb-003 has been shown to be well tolerated. This study allows the opportunity to determine if therapy with farletuzumab is effective and safe.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >18 years old
* Diagnosis of non-functional pituitary adenoma
* Able and willing to undergo surgical resection of the pituitary tumor
* Significant medical conditions must be well-controlled and stable for at least 30 days prior to signing the informed consent form

Exclusion Criteria:

* Presence of clinically significant pituitary apoplexy
* Presence of hormone-secreting adenomas
* Presence of compressive optic neuropathy due to pituitary tumor
* No prior surgical, medical, or radiation therapy in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of farletuzumab in subjects with resectable, non-functioning pituitary macroadenomas as measured by objective response in the tumor size. | Every 3 months

SECONDARY OUTCOMES:
Safety and tolerability of farletuzumab in this patient population. | Weekly for the first 3 months followed by every 2 weeks for 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wallin, MD, Study Director — Morphotek; Nelson Oyesiku, MD, PhD, FACS, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States